CLINICAL TRIAL: NCT05160662
Title: "Important Project," a Prospective Cohort Study on Pregnant Women With BMI>=35
Brief Title: The Important Project of Obese Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Karolinska Institutet
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 102030
Record Dates: First submitted 2021-11-21; First posted 2021-12-16 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Overweight and Obesity
Keywords: BMI, obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: A prospective cohort study involving all women with a BMI >35 who give birth at the women's clinic, between 2019-2023. New guidelines for this group are being developed using NICE guidelines (UK) as a model and will be tested in clinical practice
  The material will be grouped into:
  Women with BMI>=35 delivered at the hospital 2019-2020 (control group) Women with BMI>=35 delivered at the hospital 2021-2023 (where new guidelines have been used)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with BMI>=35 (2019-2020) (No Intervention): Pregnant women with BMI>=35 delivered at the hospital 2019-2020
- Women with BMI>=35 (2021-2023) (Experimental): Pregnant women with BMI>=35 delivered at the hospital 2021-2023
  Interventions: Procedure: New guidlines

INTERVENTIONS:
Procedure: New guidlines — New guidelines for this group are being developed using NICE guidelines (evidence-based recommendations for health and care in England) as a model and will be tested in clinical practice
  Arms: Women with BMI>=35 (2021-2023)

SUMMARY:
Obesity is a globally growing public health problem. In 1993, about 25% of women in Sweden were overweight (BMI over 25) or obese (BMI over 30) on the first visit to maternal health care. Twenty years later, in 2013, the corresponding proportion was 38%. Being fat increases the risk of several severe complications during pregnancy and childbirth, such as miscarriage, premature birth, congenital disabilities, intrauterine fetal death, thromboembolism, gestational diabetes, pregnancy-induced hypertension.

Purpose of the project: To assess whether the introduction of new guidelines for overweight pregnant women (BMI>35) affects the outcome of pregnancy and childbirth, such as the frequency of cesarean sections or labor inductions.

DETAILED DESCRIPTION:
A prospective cohort study involving all women with a BMI >35 who give birth at the women's clinic, Soder Hospital, Stockholm, between 2019-2023. New guidelines for this group are being developed using NICEguidelines (UK) as a model and will be tested in clinical practice.

Information from births will be collected from medical files. The information will be handled on a group basis.

Internationally, there are guidelines for how pregnancy should be handled when a woman has a high BMI. This is currently lacking in Swedish maternity care. These international guidelines have now been translated and adapted to Swedish conditions and will be tested for a 2 year period at the women's clinic.

ELIGIBILITY:
Inclusion Criteria:

* : Pregnancy where the woman has a BMI>=35 when enrolling to prenatale care

Exclusion Criteria:

* Pregnant women with BMI<35

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in unnecessary interventions | through study completion, an average of 2 years
  To assess whether the introduction of new guidelines for the group of overweight pregnant women (BMI>35) affects outcomes such as the frequency of cesareans sections or induction of labor

CONTACTS AND LOCATIONS:
Overall Officials: Eva wiberg-itzel, Principal Investigator — Karolinska Institute Sodersjukhuset Sweden
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No